CLINICAL TRIAL: NCT06223334
Title: Clinico-etiological Profile of Epileptic Syndromes in Infants and Early Childhood
Brief Title: Epileptic Syndromes in Infants and Early Childhood
Status: Recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amir Abdelaal Hasanain Abdelrahman, Assisstant Lecturer, Al-Azhar University
Other Study IDs: epilepsy syndromes
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Epileptic Syndromes
Keywords: infants; early childhood
MeSH Terms: conditions — Epileptic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- GTCS (generalized Tonic Clonic Seizures)
  Interventions: Other: No intervention
- Tonic Seizures
  Interventions: Other: No intervention
- Clonic Seizures
  Interventions: Other: No intervention
- Myoclonic Seizures
  Interventions: Other: No intervention
- Absence Seizures
  Interventions: Other: No intervention
- Focal Seizures
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — observational study to evaluate the different clinical and etiological patterns of epileptic syndromes in infants and early childhood.

SUMMARY:
To evaluate the different clinical and etiological patterns of epileptic syndromes in infants and early childhood.

DETAILED DESCRIPTION:
Epilepsy is the most common disabling neurological problem among children worldwide, and has a varying prevalence and etiological profile across the life-cycle. Onset of epilepsy prior to two-year age is more common than later in childhood.

It more commonly has a symptomatic cause and poor long-term outcome with respect to seizure-control and cognition. Previous work from India on epilepsy in infants has either focused on a single etiology, on one particular epilepsy syndrome, or on single seizure rather than epilepsy.

A recent prospective, population-based study showed an incidence of 75 per 100 000 live births prior to 6 months and 62 per 100 000 between 6 and 12 months, considerably higher than previous estimates from retrospective studies. These population-based studies are from high-resource countries, and it is noteworthy that acquired epilepsies have a higher incidence in resource-limited populations.

Traditionally, syndromes have been defined primarily by electroclinical features; however, in the last two decades, gene discovery in the epilepsies has allowed cohorts of cases with a shared genetic etiology to be studied. Consistent electroclinical phenotypes have emerged, with examples including CDKL5, MeCP2, PCDH19, STXBP1, and inv dup 15.

An epileptic syndrome is "an epileptic disorder characterised by a cluster of signs and symptoms customarily occurring together; these include such items as the type of seizure, aetiology, anatomy, precipitating factors, age of onset, severity, chronicity, diurnal and circadian cycling, and sometimes prognosis. However, in contradistinction to a disease, a syndrome does not necessarily have a common aetiology and prognosis.

An epilepsy syndrome is "a complex of signs and symptoms that define a unique epilepsy condition. This must involve more than just the seizure type; thus, for instance, frontal lobe seizures per se do not constitute a syndrome.

Furthermore, some structural, metabolic, immune, and infectious etiologies also have characteristic electroclinical phenotypes. Therefore, epilepsies due to specific genetic, structural, metabolic, immune, or infectious etiologies may also meet criteria for a syndrome, when they are associated with consistent electroclinical features and have management and prognostic implications. Epilepsies in children younger than 3-years-old can be classified by syndrome in 54% of patients and by etiology in 54%, when the latest neuroimaging, metabolic, and gene testing techniques are used. In the group younger than 12 months, etiology could be determined in 64%. By comparison, infants with severe epilepsies beginning before 18 months can be classified with an epilepsy syndrome at presentation in 64%, with the etiology being determined in 67%.

The concept of the "developmental and epileptic encephalopathy" (or DEE) recognizes that in infants presenting with severe early-onset epilepsy, neurodevelopmental comorbidity may be attributable to both the underlying cause and to the adverse effects of uncontrolled epileptic activity.

Children presenting with epilepsy very early in life experience a high burden of cognitive and behavioral comorbidity, and higher rates of drug resistance and mortality, with up to 50% showing global developmental delay 2 years after presentation. Comorbidities are more frequent among children who develop drug-resistant seizures and those with a high seizure burden.

ELIGIBILITY:
Inclusion Criteria:

For each group

* Infants and children diagnosed as epilepsy syndrome (as per International League Against Epilepsy, 2014).
* Infants and children ages ranged between 1 & 36 months.

Exclusion Criteria:

for each group

* Patients with epilepsy less than 1 month and more than 36 months.
* Patients with conditions mimic epilepsy.
* Patients with seizures related to electrolyte disturbances, inborn error of metabolism, mitochondrial diseases, white matter diseases, neurodegenerative diseases, peroxisomal disorders and non-syndromic epileptic children.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The cases will be chosen during the Child Neurology Outpatients Consults in pediatric neurology units of Al-azhar and Child Assiut University Hospitals. Based on clinical data, the patients will be divided into different epilepsy syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Epileptic syndromes in Infants and early childhood. | 2 years
  To identify the clinical profile of infants & children aged 1 to 36 mo and the characteristics of seizures in them during the Child Neurology Outpatients Consults in pediatric neurology units of Al-azhar and Child Assiut University Hospitals.
  The collected data will be statistically analyzed by statistical package for social sciences (SPSS) version 28 (IBM SPSS Inc., Chicago, US) for Windows 10. Categorical data will be expressed as numbers and percentages while continuous data will be expressed as Mean ± standard deviation (SD). The categorical variables will be compared using chi-square (χ2). The Student's T-test and ANOVA will be used for comparisons in numerical parametric data. P-value will be considered significant if < 0.05.

SECONDARY OUTCOMES:
Efficacy of treatment in epileptic syndromes in Infants and early childhood. | 2 years
  Clinical improvement will be calculated by dividing improved patients by the number of enrolled patients in each group (calculated as intended to treat and per protocol analysis). Effect size using odds ratios (with their confidence intervals, CI) of improved and not improved patients.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Abdelaal Hasanain Abdelrahman, Principal Investigator — Al-Azhar University; Emad El-Deen Mahmoud Hammad El-Daly, Study Chair — Assiut University; Mohammed Abo-Alwafa Aladawy, Study Director — Al-Azhar University
Locations (2):
- Egypt (2):
  - Assiut child university hospital, Asyut
  - AlAzhar university hospital Assiut branch, Asyut

REFERENCES:
- [Background] Scheffer IE, Berkovic S, Capovilla G, Connolly MB, French J, Guilhoto L, Hirsch E, Jain S, Mathern GW, Moshe SL, Nordli DR, Perucca E, Tomson T, Wiebe S, Zhang YH, Zuberi SM. ILAE classification of the epilepsies: Position paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):512-521. doi: 10.1111/epi.13709. Epub 2017 Mar 8. PMID 28276062
- [Background] Farghaly WM, Abd Elhamed MA, Hassan EM, Soliman WT, Yhia MA, Hamdy NA. Prevalence of childhood and adolescence epilepsy in Upper Egypt (desert areas). Egypt J Neurol Psychiatr Neurosurg. 2018;54(1):34. doi: 10.1186/s41983-018-0032-0. Epub 2018 Nov 9. PMID 30532513
- [Background] Howell KB, Freeman JL, Mackay MT, Fahey MC, Archer J, Berkovic SF, Chan E, Dabscheck G, Eggers S, Hayman M, Holberton J, Hunt RW, Jacobs SE, Kornberg AJ, Leventer RJ, Mandelstam S, McMahon JM, Mefford HC, Panetta J, Riseley J, Rodriguez-Casero V, Ryan MM, Schneider AL, Smith LJ, Stark Z, Wong F, Yiu EM, Scheffer IE, Harvey AS. The severe epilepsy syndromes of infancy: A population-based study. Epilepsia. 2021 Feb;62(2):358-370. doi: 10.1111/epi.16810. Epub 2021 Jan 21. PMID 33475165
- [Background] Kharod P, Mishra D, Juneja M. Drug-resistant epilepsy in Indian children at a tertiary-care public hospital. Childs Nerv Syst. 2019 May;35(5):775-778. doi: 10.1007/s00381-019-04084-5. Epub 2019 Feb 13. PMID 30758667
- [Background] Kolc KL, Sadleir LG, Scheffer IE, Ivancevic A, Roberts R, Pham DH, Gecz J. A systematic review and meta-analysis of 271 PCDH19-variant individuals identifies psychiatric comorbidities, and association of seizure onset and disease severity. Mol Psychiatry. 2019 Feb;24(2):241-251. doi: 10.1038/s41380-018-0066-9. Epub 2018 Jun 11. PMID 29892053
- [Background] Symonds JD, Elliott KS, Shetty J, Armstrong M, Brunklaus A, Cutcutache I, Diver LA, Dorris L, Gardiner S, Jollands A, Joss S, Kirkpatrick M, McLellan A, MacLeod S, O'Regan M, Page M, Pilley E, Pilz DT, Stephen E, Stewart K, Ashrafian H, Knight JC, Zuberi SM. Early childhood epilepsies: epidemiology, classification, aetiology, and socio-economic determinants. Brain. 2021 Oct 22;144(9):2879-2891. doi: 10.1093/brain/awab162. PMID 34687210